CLINICAL TRIAL: NCT06370156
Title: Evaluation of TWEAK in Plaque Psoriasis and Psoriatic Arthritis Patients Treated With Adalimumab and Methotrexate: Case Control Study
Brief Title: Evaluation of TWEAK in Plaque Psoriasis and Psoriatic Arthritis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Other Study IDs: TWEAK in plaque psoriasis
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A : (Adalimumab therapy): About 30 patients suffering from Plaque Psoriasis and will take Adalimumab therapy orally.
  Correlation between serum& TWEAK levels and Psoriasis Area and Severity Index (PASI) score and the ACR score pre and post Adalimumab therapy
  Interventions: Drug: Adalimumab
- Group B : (methotrexate therapy): About 30 patients suffering from Psoriatic arthritis and will take methotrexate therapy orally.
  Correlation between serum& TWEAK levels and Psoriasis Area and Severity Index (PASI) score and the ACR score pre and post methotrexate therapy
  Interventions: Drug: Adalimumab
- Group C: (control Group):: About 40 healthy individuals selected as control group as related to age, sex ,BMI matching with healthy individuals
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — To suggests the role of TWEAK and the effectiveness of different treatments like adalimumab and methotrexate in managing plaque psoriasis and psoriatic arthritis.
  Other Names: Methotrexate

SUMMARY:
Psoriasis vulgaris is associated with significant comorbidity including depression, increased risk of cardiovascular events, diminished quality of life, as well as overall increased mortality.

Moreover, concomitant psoriatic arthritis is present in up to 40% of psoriasis patients or will develop in the future.

To enhance quality of life and potentially lower the risk of concomitant disease in psoriasis patients, effective treatment of this immune-mediated systemic inflammatory disease is required

DETAILED DESCRIPTION:
Psoriasis vulgaris is associated with significant comorbidity including depression, increased risk of cardiovascular events, diminished quality of life, as well as overall increased mortality.

The cytokine tumor necrosis factor (TNF)-related weak inducer of apoptosis (TWEAK), in cooperation with its sole receptor, Fn14, is involved in miscellaneous biological and pathological processes .

The main role of TWEAK is in the induction of pro-inflammatory cytokines and chemokines. The upregulation of TWEAK and Fn14 occurs in many human skin disorders, including cutaneous lupus erythematosus, bullous pemphigoid, and dermatomyositis . There is a lack of studies examining the role of TWEAK in patients with psoriasis or psoriatic arthritis.

The introduction of anti-tumor necrosis factor-α inhibitors (anti-TNF agents) has significantly improved outcomes among patients with PsA but a proportion of patients have an inadequate response or poor tolerability to these agents.

Adalimumab treatment continuation in routine clinical practice may lead to benefits for remission and low disease activity among patients with psoriasis, psoriatic arthritis, or axial spondyloarthritis who did not achieve their treatment goals at 12 weeks, according to recent findings.

Methotrexate (MTX)was approved for the treatment of psoriasis by the US Food and Drug Administration (FDA). At present, the drug is indicated for the treatment of practically all forms of moderate or severe psoriasis, including psoriatic arthritis .

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with psoriasis vulgaris and Psoriatic arthritis.
* Active PsA with three or more tender and swollen joints and met the CASPAR, despite previous treatment with NSAIDs, DMARDs or anti-TNFs

Exclusion Criteria:

* Previously received biologic immunomodulating agents, except for those targeting TNF
* Previously been treated with three or more different TNF inhibitors
* Active, ongoing inflammatory diseases other than PsA
* Active TB (patients with latent TB had to commence treatment for latent TB before study entry)
* A history of hepatitis B or C, human immunodeficiency virus, or any active systemic infection within the 2 weeks before baseline
* History of ongoing, chronic or recurrent infections, or evidence of active TB infection
* History of malignancy within the past 5 years (except for basal cell carcinoma or actinic keratosis that has been treated with no evidence of recurrence in the past 3 months, in situ cervical cancer or non-invasive malignant colon polyps that had been removed)
* Underlying metabolic, hematological, renal, hepatic, pulmonary, neurological, endocrine, cardiac, infectious or gastrointestinal conditions which, in the opinion of the investigator, immunocomprimised the patient and/or placed the patient at unacceptable risk for participation
* Pregnant or nursing (lactating) women and women of child-bearing potential unwilling to use effective contraception during the study and for 16 weeks after stopping treatment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * TWEAK serum level assessment: blood sample (about 5cc) from the antecubital vessel of well-being control candidates and psoriatic candidates before and after MTX and Adalimumab therapy.
  * Lipid profile will be calculated for patients treated, Liver & renal function will be measured and HCV, HBV and TB .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Treatment of psoriasis vulgaris and psoriatic arthritis | 1 year
  to see the efficacy of drug study in improving the prognosis of patients with psoriasis vulgaris and psoriatic arthritis.

SECONDARY OUTCOMES:
Evaluation of serum TWEAK | 1 year
  To detect the correlation between serum TWEAK the PASI score and the ACR score pre and post Methotrexate and Adalimumab therapy

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley Hospitals, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided